CLINICAL TRIAL: NCT03962816
Title: A Prospective Study on the Immunogenicity and Persistence of Hepatitis B Vaccine in Methadone Maintenance Treatment Patients
Brief Title: Immunogenicity and Persistence of Hepatitis B Vaccination in Methadone Maintenance Treatment Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanxi Medical University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Suping Wang, Professor, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018ZX10721202001002002
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B Vaccine; Randomized Controlled Trial; Methadone Maintenance Treatment Patients; Immunogenicity; Long-term Immune Response
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 µg at months 0, 1, and 6 (Experimental): 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, and 6
- 20 µg at months 0, 1, 2,and 6 (Experimental): 20 µg recombinant hepatitis B vaccine with four injections at months 0, 1, 2, and 6
  Interventions: Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6
- 60 µg at months 0, 1, 2,and 6 (Experimental): 60 µg recombinant hepatitis B vaccine with four injections at months 0, 1, 2, and 6
  Interventions: Biological: 60 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6

INTERVENTIONS:
Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, and 6 — three-dose, 20 µg per dose
  Arms: 20 µg at months 0, 1, and 6
Biological: 20 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6 — four-dose, 20 µg per dose
  Arms: 20 µg at months 0, 1, 2,and 6
Biological: 60 µg recombinant hepatitis B vaccine at months 0, 1, 2, and 6 — four-dose, 60 µg per dose
  Arms: 60 µg at months 0, 1, 2,and 6

SUMMARY:
At present, Methadone Maintenance Treatment Patients of Hepatitis B Vaccination in are vaccinated with hepatitis B vaccine according to the standard three-dose schedule immunization program, and the effect of preventing HBV infection is not ideal.

This is a randomized, controlled trial. The study will evaluate the immunogenicity and persistence of 20 µg and 60 µg recombinant hepatitis B vaccine with three or four injections at months 0, 1, and 6 or 0, 1,2, and 6 in Methadone Maintenance Treatment Patients

DETAILED DESCRIPTION:
Participants are randomized in a ratio of 1:1:1 into 20 µg recombinant hepatitis B vaccine group at months 0, 1, and 6 or 20µg recombinant hepatitis B vaccine group at months 0, 1, 2, and 6 or 60µg recombinant hepatitis B vaccine group at months 0, 1, 2, and 6. HBsAg and anti-HBs will be tested during the study period. Adverse reactions will be recorded after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Serologically negative for hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs) and hepatitis B core antibody (anti-HBc) at enrollment
* Sign informed consent, willing to participate in this study

Exclusion Criteria:

* Being pregnant
* Intolerance or allergy to any component of the vaccine
* Any vaccination during the month preceding enrollment
* Patients with severe acute or chronic diseases (such as liver disease, blood disease, cancer), acute onset of chronic diseases and fever
* Patient with HIV Infection
* The use of immunosuppressive agents in patients with nearly three months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-26 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anti-HBs Seroconversion Rate at Month 7 | Month 7
  Anti-HBs Seroconversion Rate at month 7 as measured by CMIA

SECONDARY OUTCOMES:
Anti-HBs concentration at month 7 | Month 7
  Anti-HBs concentration at month 7 as measured by CMIA
Occurrence of Adverse Events After Vaccination | Within 7 days after the vaccination
  Occurrence of adverse reactions within 7 days after vaccination with the hepatitis
Anti-HBs Seroconversion Rate at month 12 | Month 12
  Anti-HBs Seroconversion Rate at month 12 as measured by CMIA
Anti-HBs concentration at month 12 | Month 12
  Anti-HBs concentration at month 12 as measured by CMIA
Anti-HBs Seroconversion Rate at month 18 | Month 18
  Anti-HBs Seroconversion Rate at month 18 as measured by CMIA
Anti-HBs concentration at month 18 | Month 18
  Anti-HBs concentration at month 18 as measured by CMIA
Anti-HBs Seroconversion Rate at month 30 | Month 30
  Anti-HBs Seroconversion Rate at month 30 as measured by CMIA
Anti-HBs concentration at month 30 | Month 30
  Anti-HBs concentration at month 30 as measured by CMIA
Anti-HBs Seroconversion Rate at month 42 | Month 42
  Anti-HBs Seroconversion Rate at month 42 as measured by CMIA
Anti-HBs concentration at month 42 | Month 42
  Anti-HBs concentration at month 42 as measured by CMIA

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, PhD, Principal Investigator — Shanxi Medical University
Locations (1):
- Xinghualing Methadone Drug Point, Taiyuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mo X, Men Z, Gao L, Gao Y, Yao T, Liu Y, Yuan Y, Xue T, Wang F, Wang S, Wang K, Liang X, Feng Y. Immunogenicity persistence after four intramuscular triple-dose or standard-dose hepatitis B vaccine in patients receiving methadone maintenance treatment: A 1-year follow-up study in China. Hum Vaccin Immunother. 2025 Dec;21(1):2447108. doi: 10.1080/21645515.2024.2447108. Epub 2025 Jan 17. PMID 39819251
- [Derived] Feng Y, Yao T, Gao Y, Li H, Dong S, Wu Y, Liu Y, Li J, Liu C, Liu J, Xue T, Yuan Y, Wu J, Wang F, Liang X, Wang S. Immunogenicity, safety, and compliance of high- and standard-strength four-dose hepatitis B vaccination regimens in patients receiving methadone maintenance therapy in China: a randomized, parallel-arm controlled trial. Expert Rev Vaccines. 2021 Dec;20(12):1629-1635. doi: 10.1080/14760584.2021.1977629. Epub 2021 Sep 16. PMID 34503367